CLINICAL TRIAL: NCT05817149
Title: Perioperative Examination of Inflammatory Markers in Relation to Sentinel Lymph Node Biopsy in Patients With Melanoma; a Pilot Study
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Karoline Assifuah Kristjansen, MD, Ph.d-student, Aalborg University Hospital
Other Study IDs: 2021-050
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Melanoma; Surgery
Keywords: Melanoma; Surgery; Neutrophil-to-lymphocyte ratio; Surgical inflammation
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Perioperative blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with melanoma: Patients with melanoma undergoing sentinel lymph node biopsy with perioperative blood samples.
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — Blood samples

SUMMARY:
We want to test if an association between sentinel lymph node biopsy (SLBN) and a systemic inflammatory response can be made.

DETAILED DESCRIPTION:
Sentinel lymph node biopsy (SLBN) is essential in staging melanoma and properly selecting patients for adjuvant immunotherapy. However, surgically induced inflammation can potentially aid in progression of remaining malignant cells and affect prognosis. The inflammatory marker neutrophil-to-lymphocyte ratio (NLR) is also a negative prognostic and predictive marker in serval malignancies, among melanoma. However, it is not yet established if SLNB induces a systemic inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years of age)
* Diagnosed with invasive cutaneous melanoma
* Eligible for SLNB (Melanoma stage ≥ T1b)
* Obtained signed informed consent

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (n=20) diagnosed with malignant melanoma and scheduled for SLNB at Aalborg University Hospital were consecutively included from June 2021 to October 2021.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Neutrophil-to-lymphocyte ratio | 1 Day
  Ratio between neutrophil granulocytes and lymphocytes

SECONDARY OUTCOMES:
Pro-inflammatory cytokines | 1 Day
  IL-1b, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, and IFN-γ
Acute phase reactants | 1 Day
  CRP, LDH

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, The North Denmark Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided